CLINICAL TRIAL: NCT00961987
Title: Innovation to the Provision of Maternity Care in Hamilton: An Inter- and Intraprofessional Collaboration
Brief Title: Innovation to Providing Interprofessional Maternity Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McMaster University (Other)
Responsible Party: Dr. Keyna Bracken, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05-1309
Record Dates: First submitted 2009-08-18; First posted 2009-08-19 (Estimated); Last update posted 2009-08-19 (Estimated); Status verified 2009-08

CONDITIONS: Pregnancy
Keywords: Maternity care; Interprofessional collaboration; Continuity of Care; Integration

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Collaborative model (Experimental): Patients will be referred (if necessary) to an obstetrician who will be co-located in the Maternity Centre and who will be part of the collaborative model of maternity care.
  Interventions: Other: Collaborative model
- Usual care (Active Comparator): At present, if Maternity Centre patients require the specialized services of an obstetrician, the current standard of care is to refer them to obstetricians located offsite with no professional ties to the Maternity Centre
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Collaborative model — Patients will be referred (if necessary) to an obstetrician who will be co-located in the Maternity Centre and who will be part of the collaborative model of maternity care.
  Arms: Collaborative model
Other: Usual care — At present, if Maternity Centre patients require the specialized services of an obstetrician, the current standard of care is to refer them to obstetricians located offsite with no professional ties to the Maternity Centre
  Arms: Usual care

SUMMARY:
The aim of this pilot project is to determine if there are differences in patient outcomes and healthcare utilization between patients randomly assigned to usual care (a collaborative model of maternity care with co-located healthcare professionals but with referrals to off-site obstetricians) or to a collaborative model of maternity care with co-located healthcare professionals, including obstetricians. It is hypothesized that by creating a seamless interface between obstetrical consultation and ongoing longitudinal maternity care, patient outcomes (birth outcome data), patient satisfaction and healthcare utilization, including number of outpatient visits, ultrasounds, laboratory tests, consultations, etc, will be improved in the intervention group compared with the group receiving usual care. The results could potentially lead to other sites adopting this innovative model of maternity healthcare delivery.

ELIGIBILITY:
Inclusion Criteria:

* 16 years of age or older
* Attending their intake appointment at the Centre
* Ability to understand English
* Legal status in Canada

Exclusion Criteria:

-

Ages: 16 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 700 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Patient outcomes (birth outcomes) | 9 months

SECONDARY OUTCOMES:
Patient satisfaction | 9 months
Healthcare utilization | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Keyna Bracken, MD, Principal Investigator — McMaster University
Locations (1):
- Maternity Centre, Hamilton, Ontario, Canada